CLINICAL TRIAL: NCT06260930
Title: Role od Chest Ultrasonography in Interstitial Lung Diseases
Brief Title: Value of Chest Ultrasonography in ILD Screening
Status: Completed | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Shazly Ahmed, Associate professor, Aswan University
Other Study IDs: Value of chest ultrasonography
Record Dates: First submitted 2024-01-09; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main aim of this study is to detect the value of transthoracic ultrasonography in the diagnosis and assessment of ILDs in correlation to chest X- ray, blood gases, pulmonary function test and echocardiography and to compare it with high resolution CT (HRCT) as a golden diagnostic investigation.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) refers to a group of disorders that are characterized by varying combinations of inflammation and fibrosis involving the space between the epithelial and endothelial basement membranes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) diagnosed with ILD
* All patients must fulfil the 2018 criteria for HRCT chest finding for the diagnosis of Usual interstitial pneumonia (UIP) form

Exclusion Criteria:

* Patients with cardiac diseases (Left-sided Heart failure, pulmonary edema) [they may have findings of multiple B lines on transthoracic ultrasound examination which mimic ILD findings].
* Patients with chronic kidney diseases (as patients presented with nephrogenic pulmonary edema may have findings of multiple B lines on transthoracic ultrasound examination which mimic ILD findings).

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be recruited from the Department of Chest, Aswan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the lung sonography for interstitial lung disease screening | 12 months
  To estimate the sensitivity and specificity of the lung sonography for interstitial disease screening in comparison with HRCT. [Time Frame: 12 months]

REFERENCES:
- [Background] Deconinck B, Verschakelen J, Coolen J, Verbeken E, Verleden G, Wuyts W. Diagnostic workup for diffuse parenchymal lung disease: schematic flowchart, literature review, and pitfalls. Lung. 2013 Feb;191(1):19-25. doi: 10.1007/s00408-012-9433-5. Epub 2012 Nov 13. PMID 23149802